CLINICAL TRIAL: NCT00673647
Title: Evaluation of the Cognitive-behavioral Treatment Programme CANDIS in the German Outpatient Treatment Service System (CANDIS-II)
Brief Title: CANDIS-II: Evaluation of the Cognitive-behavioral Treatment Programme CANDIS
Acronym: CANDIS-II
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Technische Universität Dresden (Other)
Collaborators: Federal Ministry of Health (Ambiguous)
Responsible Party: PhD Eva Hoch, Technische Universitaet Dresden
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IIA5-2507DSM407
Record Dates: First submitted 2008-05-01; First posted 2008-05-07 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Cannabis Use Disorders
Keywords: cannabis; dependence; marijuana; CBT; efficacy of CBT for cannabis use disorders
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Individual psychotherapy including cognitive behavioral components, motivational interviewing techniques and case management
  Interventions: Behavioral: Cognitive-behavioral treatment
- 2 (No Intervention): Delayed treatment control group

INTERVENTIONS:
Behavioral: Cognitive-behavioral treatment — 10 sessions of individual psychotherapy including cognitive-behavioral treatment, motivational enhancement and a psychosocial problem training.
  Other Names: delayed treatment control group
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the cognitive-behavioral treatment program CANDIS among n=450 patients with cannabis use disorders in a mulicenter randomized-controlled clinical trial (n=11 outpatient treatment centers).

ELIGIBILITY:
Inclusion Criteria:

* motivation to change cannabis use
* age 16 or older
* current (12 mth) regular cannabis use (at least 2 days a week)
* informed consent to the study procedures and assessments

Exclusion Criteria:

* current alcohol or any illicit drug dependence syndrome according to DSM-IV other than due to cannabis
* lifetime history of any psychotic disorder
* current severe episode of Major depression
* current panic-agoraphobic disorder (severe)
* severe learning disability, brain damage or pervasive developmental disorder
* currently acute suicidality
* not fluent in german language
* any other current treatment for cannabis use disorders

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
abstinence, defined as no evidence of cannabis use during the past 4 weeks as evidenced by self report and a negative urine screen; number of times a cannabis product was used in the past 4 weeks; retention rate | at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Ulrich Wittchen, PhD, Study Director — Technische Universitaet Dresden; Gerhard Buehringer, PhD, Study Director — Technische Universitaet Dresden; Eva Hoch, PhD, Principal Investigator — Technische Universitaet Dresden
Locations (11):
- Germany (11):
  - Psychosoziale Beratungs- und Behandlungsstelle für Suchtgefährdete und -kranke, Bautzen
  - LogIn Jugend- und Suchtberatung, Berlin
  - Therapieladen e.V., Berlin
  - Jugend- und Drogenberatung Braunschweig, Braunschweig
  - Jugend- und Drogenberatung Dresden, Dresden
  - Die Boje - Suchtberatung und Behandlung, Hamburg
  - Drobs Hannover, Hanover
  - Caritas-Fachambulanz für junge Suchtkranke, München
  - Suchtambulanz der LWL-Klinik Münster, Münster
  - Caritas Fachambulanz für Suchtprävention und Rehabilitation Osnabrück, Osnabrück
  - Release Stuttgart e.V. & Ambulante Beratungs- und Behandlungsstelle Klinikum Stuttgart, Stuttgart

REFERENCES:
- [Derived] Hoch E, Buhringer G, Pixa A, Dittmer K, Henker J, Seifert A, Wittchen HU. CANDIS treatment program for cannabis use disorders: findings from a randomized multi-site translational trial. Drug Alcohol Depend. 2014 Jan 1;134:185-193. doi: 10.1016/j.drugalcdep.2013.09.028. Epub 2013 Oct 8. PMID 24176199
- See also: Related Info — http://www.candis-projekt.de
- See also: Related Info — http://www.psychologie.tu-dresden.de